CLINICAL TRIAL: NCT03049332
Title: Self- and Family-management Intervention in HIV+ Chinese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Beijing Ditan Hospital (Other); Shanghai Public Health Clinical Center (Other Government); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1207010522; K23NR014107-02 (NIH)
Record Dates: First submitted 2017-02-07; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Hiv
Keywords: Quality of Life
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The same group of individuals will be measured pre and post intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): HIV+ Chinese women in China and a family member will be recruited for the pilot testing of the intervention.
  Interventions: Behavioral: self- and family-management intervention sessions

INTERVENTIONS:
Behavioral: self- and family-management intervention sessions — The self- and family management intervention will have six elements: (a) biofeedback for relaxation; (b) family support; (c) coping skills; (d) anxiety, stress, and depression management; (e) cognitive-behavioral management skills; and (f) psycho-educational classes.

SUMMARY:
This project is to develop a culturally sensitive and feasible self- and family-management intervention that will assist HIV+ Chinese women and their families to manage the illness and improve quality of life and clinical outcomes.

DETAILED DESCRIPTION:
The study will be conducted in 3 phases.

Phase 1: The PI conducted a secondary qualitative analysis of in-depth interviews to further illuminate the sociocultural and family context of HIV+ Chinese women. The data were obtained from three previous projects conducted in China from 2005 to 2011.

Phase 2: The PI developed and adapted a theory-driven, culturally sensitive and feasible intervention to improve the quality of life and clinical outcomes of HIV+ Chinese women and their families.

Phase 3: The PI conducted a feasibility, compliance, and acceptability study for a self- and family-management intervention with HIV+ women and of their family members.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for HIV+ women.

* be at least 18 years of age,
* be able to give informed consent for the study and to cognitively participate,
* be receiving clinical care at Ditan Hospital and SPHCC,
* have been diagnosed with HIV within the past 12 months,
* have disclosed their status to at least one family member and willing to invite that family member to the intervention,
* be well enough to attend counseling sessions at the hospital, and
* be able to attend follow-up visits at the hospital.

Inclusion criteria for family members.

* be 18 years of age,
* be able to give informed consent for the study and to cognitively participate,
* have a female family member who is HIV+, and is currently receiving clinical care at Ditan Hospital and SPHCC,
* be a family member who are taking care of the female HIV+ family member,
* be well enough to attend counseling sessions at the hospital, and
* be able to attend follow-up visits at the hospital.

Exclusion Criteria:

Exclusion criteria for HIV+ women

* history of an affective illness such as depression or bipolar disease,
* are under age 18, or
* are unwilling or unable to bring a family member to participate in the study.

Exclusion criteria for family members.

* have a history of an affective illness such as depression or bipolar disease,
* are under age 18,
* or are unwilling or unable to come with their HIV+ family member to participate the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
retention rates | 6 months
  the percentage of self- and family-management intervention sessions attended by both HIV+ women and one family member
compliance with data collection procedures | 6 months
  includes attending counseling sessions and completing questionnaires
acceptability | 6 months
  including reports of burden related to the study and/or intervention procedures measured by intervention session logs and exit interview
feelings of safety | 6 months
  family members and study participants feelings of safety related to participating in this project measured by intervention session logs and exit interview

CONTACTS AND LOCATIONS:
Overall Officials: Weiti Chen, Principal Investigator — Yale University School of Nursing
Locations (2):
- China (2):
  - Beijing Ditan Hospital, Beijing
  - Shanghai Public Health Clinical Center, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen WT, Shiu C, Zhang L, Zhao H. Care engagement with healthcare providers and symptom management self-efficacy in women living with HIV in China: secondary analysis of an intervention study. BMC Public Health. 2022 Jun 15;22(1):1195. doi: 10.1186/s12889-022-13573-3. PMID 35705934